CLINICAL TRIAL: NCT04020783
Title: A Prospective Study of the Incidence and Outcomes of Primary Aldosteronism in Chinese Hypertensive Patients
Brief Title: Primary Aldosteronism: Prospective Screening Registry in China
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Chinapaps
Record Dates: First submitted 2019-06-26; First posted 2019-07-16 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Primary Aldosteronism
Keywords: Primary aldosteronism; Screening
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: sequential
  Interventions: Other: NO Intervention

INTERVENTIONS:
Other: NO Intervention — NO Intervention

SUMMARY:
1. Study name: A prospective study of the incidence and outcomes of Primary aldosteronism in Chinese hypertensive patients
2. Rationale: Unlike essential hypertension, secondary hypertension is caused by certain defined diseases or causes. For this reason, secondary hypertension can often be cured or effectively controlled. As one of the most common types of secondary hypertension, it is estimated that primary aldosteronism (PA) accounts for 5%-10% of all hypertensive patients, accounting for about 20% of patients with refractory hypertension.
3. Objective: 1) Collect and analyze the population and disease characteristics of Chinese PA patients; 2) Strengthen the awareness of screening for PA in people with high blood pressure.
4. Study design: Prospective , multi-center, observational study.
5. Study population: Hypertensive patients with high suspected or confirmed of primary aldosteronism.
6. Treatment: Standardized diagnosis and treatment procedure as recommended in the international guidelines of PA.
7. Follow up: 6, 12 and 24 months after diagnosis.
8. Sample size estimation: About 10 thousand.
9. Timeline: Start of subjects enrollment: July 2019; End of subjects enrollment: December 2022; End of study: December 2024.
10. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

DETAILED DESCRIPTION:
1. Study name: A prospective study of the incidence and outcomes of Primary aldosteronism in Chinese hypertensive patients
2. Rationale: Hypertension is the most common cardiovascular disease, a serious cardiovascular disease state, and the most important risk factor for serious cardiovascular and cerebrovascular complications such as stroke, myocardial infarction, heart failure, and renal insufficiency. The China Cardiovascular Disease Report 2018 pointed out that the total number of people suffering from hypertension in China reached 245 million, which has become a major public health problem affecting people's health and restricting economic development.

   Unlike essential hypertension, secondary hypertension is caused by certain defined diseases or causes. For this reason, secondary hypertension can often be cured or effectively controlled with the appropriate treatment. As one of the most common types of secondary hypertension, it is estimated that primary aldosteronism (PA) accounts for 5%-10% of all hypertensive patients, accounting for about 20% of patients with refractory hypertension. Therefore, how to find out patients with PA in hypertensive population in time and carry out targeted treatment is a challenge that cardiovascular professional clinicians must face.

   Diagnostic PA begins with screening. With the advancement of detection technology, especially the clinical popularity of chemiluminescence detection of plasma aldosterone and renin concentration, the detection of suspected PA patients by plasma aldosterone renin ratio (ARR) in medium-sized hospitals has become a reality. Due to the limitations of clinical examination, there are only a few hospitals that can actually perform the etiological diagnosis of PA. As long as we can screen out suspected PA patients, it is a major advancement in the diagnosis and treatment of secondary hypertension. In order to popularize the clinical application of PA screening and diagnosis technology, systematically collect clinical data of PA patients in China, it is necessary to carry out PA screening registration research in hypertensive patients.
3. Objective: 1) Collect and analyze the population and disease characteristics of Chinese PA patients; 2) Strengthen the awareness of screening for PA in people with high blood pressure.
4. Study design: Prospective, multi-center observational study.
5. Study population: Hypertensive patients with high suspected or confirmed of primary aldosteronism. High suspected of primary aldosteronism include 6 types of hypertensive patients: 1) persistent blood pressure > 160/100 mmHg, refractory hypertension ( combined with 3 antihypertensive drugs, including diuretics, blood pressure > 140/90 mmHg), Combined use of 4 or more antihypertensive drugs, blood pressure <140/90 mmHg; 2) hypertension combined with spontaneous or diuretic hypokalemia; 3) hypertension with adrenalaccidental tumor; 4) family history of early onset hypertension Or hypertensive patients with a family history of cerebrovascular accidents (<40 years old); 5) first-degree relatives with hypertension in patients with primary aldosteronism; 6) hypertension with obstructive respiratory sleep apnea. The other study population is the PA patients confirmed.
6. Treatment: Standardized diagnosis and treatment procedure as recommended in the international guidelines of PA. Hypertensive Patients should adjust antihypertensive medication before ARR testing to ensure accurate ARR measurements. Patients with positive ARR results (more than 40) are suspected PA and need confirmation test, such as Saline infusion test or Captopril test. PA patients should undergo a sub-type diagnosis, such as adrenal CT, AVS. Patients with PA confirmed are treated with drugs or surgery after diagnosis.
7. Follow up: 6, 12 and 24 months after diagnosis.
8. Sample size estimation: About 10 thousand.
9. Timeline: Start of subjects enrollment: July 2019; End of subjects enrollment: December 2022; End of study: December 2024.
10. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Eligibility criteria

1. Age: more than or equal to 18 years old;
2. Hypertensive patients ;
3. ARR > 40;
4. Informed consent;

Exclusion criteria:

Not eligible for inclusion or in situations considered unqualified for the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients with high suspected or confirmed of PA. High suspected of PA include 6 types of hypertensive patients: 1) persistent blood pressure > 160/100 mmHg, refractory hypertension ( combined with 3 antihypertensive drugs, including diuretics, blood pressure > 140/90 mmHg), Combined use of 4 or more antihypertensive drugs, blood pressure <140/90 mmHg; 2) hypertension combined with spontaneous or diuretic hypokalemia; 3) hypertension with adrenalaccidental tumor; 4) family history of early onset hypertension or hypertensive patients with a family history of cerebrovascular accidents (<40 years old); 5)first-degree relatives with hypertension in patients with PA; 6) hypertension with obstructive respiratory sleep apnea. The other study population is the PA patients confirmed.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ARR positive rate | 1 day
  ARR positive rate in the high suspicion of PA.
PA confirmed diagnostic rate | 1 month
  The rate of PA confirmed diagnosis in highly suspected PA population.
The change of office blood pressure | 24 months
  Comparison of blood pressure between baseline and 6/12/24 months.
The rate of incidence of cardiovascular events | 24 months
  The rate of incidence of cardiovascular events in the PA patients,such as cerebral infarction, hypertensive nephropathy, myocardial infarction and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, MD, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided